CLINICAL TRIAL: NCT01390051
Title: Can Treatment With Low Molecular Weight Heparin During Pregnancy With Intrauterine Growth Restriction Increase Birth Weight?
Brief Title: Can Low Molecular Weight Heparin During Pregnancy With Intrauterine Growth Restriction Increase Birth Weight?
Acronym: IUGR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-20110042
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: Fetal Growth Retardation
Keywords: birth weight; thrombosis; anticoagulant therapy
MeSH Terms: conditions — Fetal Growth Retardation; Birth Weight; Thrombosis | interventions — Tinzaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Innohep (Active Comparator): Tinzaparin 4500 I.U. sub cutaneous once daily until gestational week 37
  Interventions: Drug: Innohep (Tinzaparin); Drug: tinzaparin
- no treatment (No Intervention)

INTERVENTIONS:
Drug: Innohep (Tinzaparin) — Dose: 4,500 IU daily in half of the study populationrandomised to treatment
  Other Names: Innohep
  Arms: Innohep
Drug: tinzaparin — Dose 4,500 IE daily
  Other Names: Innohep
  Arms: Innohep

SUMMARY:
The purpose of the study is to investigate if treatment with an anticoagulant drug increases birth weight in pregnancies complicated by fetal growth restriction.

DETAILED DESCRIPTION:
Clinical purpose:

1. To examine whether treatment with low molecular weight heparin in pregnant women with Intrauterine Growth Restriction (IUGR)increases the birth weight of the child. Our hypothesis is that an increased birth weight leads to reduced morbidity and mortality among these children.

Laboratory purposes:

1. To evaluate three new methods to monitor the effect of LMWH.
2. To investigate if 2 biochemical markers are positive predictors of IUGR IUGR is defined as a foetus that grows less than expected. IUGR is estimated to occur in up to 5% of all pregnancies, and IUGR is the second most common cause of perinatal morbidity and mortality. Thus, 75% of all stillbirths are caused by IUGR. IUGR is diagnosed by ultrasonography. In IUGR the uteroplacental blood flow is often compromised resulting in foetal growth restriction.

Design: The study is a prospective randomised study where pregnant women with suspected severe IUGR are randomised either to treatment with Innohep® or no treatment. Half of the women receive Innohep® and half of the women do not receive treatment.

Endpoints The primary endpoint is the difference in birth weight in children born of women receiving Innohep® during pregnancy and children born of women who have not received Innohep® during pregnancy

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy
2. IUGR shown by ultrasonography:
3. Can understand and read Danish

Exclusion Criteria:

1. Age below 18 years
2. Pregestational weight < 90 kilograms
3. Not able to give informed consent
4. Chronic kidney disease with creatinine >150 μmol/l
5. Chronic hypertension with blood pressure >140/90 mmHg
6. Diabetes mellitus; type 1 or 2 or gestational diabetes
7. Inflammatory bowel disease
8. Severe heart disease (including mechanical heart valves)
9. Drug or alcohol abuse
10. Known coagulopathy (von Willebrand disease, thrombocytopenia, carrier of haemophilia)
11. Treatment with vitamin K antagonists
12. Known allergy to low LMWH
13. Previous heparin-induced thrombocytopenia (HIT (type II))
14. Clinically significant bleeding within the last month
15. Women with indication for prophylactic treatment with LMWH during pregnancy e.g. previous thromboembolic disease or serious types of thrombophilia (deficiency of antithrombin, protein C or protein S)
16. Chromosome anomaly in the child
17. Severe malformations in the child
18. Contraindication to Innohep®
19. Gestational week > 32 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
birth weight | Birth weight registered at birth
  We compare birth weight in children born of women from the 2 study arms

SECONDARY OUTCOMES:
maternal morbidity | Comorbidity registered up to one year after birth

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Mette Hvas, PhD, professor, Principal Investigator — Department of Clinical Biochemistry, Aarhus University Hospital, Denmark
Locations (3):
- Denmark (3):
  - Consultant phD professor Anne-Mette Hvas, Aarhus, Central Jutland
  - Department of Obstetrics, Herning
  - Department of Obstetrics, Randers